CLINICAL TRIAL: NCT05552001
Title: ISIdE: Open Label, Multicentric, Single-arm Phase IIIB Trial to Evaluate the Safety and Efficacy of Sacituzumab Govitecan in Triple Negative Metastatic Breast Cancer Patients With a Biomarker Analysis
Brief Title: Safety and Efficacy Analysis of an Antibody Associated With a Chemotherapy for Patients With a Triple Negative Metastatic Breast Cancer
Acronym: ISIdE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC-BCG-2204; 2022-502369-10-00 (Other: EU CT Number)
Record Dates: First submitted 2022-09-20; First posted 2022-09-23 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Triple Negative Breast Cancer; Metastatic Breast Cancer
Keywords: breast cancer; metastatic; triple negative; sacituzumab govitecan; biomarker analysis
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms; Neoplasm Metastasis | interventions — sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm receiving sacituzumab govitecan (Experimental)
  Interventions: Drug: Sacituzumab govitecan

INTERVENTIONS:
Drug: Sacituzumab govitecan — Sacituzumab Govitecan (SG) is given by intervenous route, 10 mg/kg on day 1 and day 8 of 21-day treatment cycles. Patient will receive treatment until disease progression, unacceptable toxicity, or decision to withdraw its participation.
  Other Names: trodelvy

SUMMARY:
ISIdE is an European, multicentric study that aims to assess the efficacy of Sacituzumab Govitecan (SG) in locally advanced or metastatic triple-negative breast cancer where the disease has progressed despite chemotherapy or within 6 months after the end of curative treatments in order to:

1. evaluate the treatment efficacy in less pretreated patients.
2. identify biomarkers that could predict response or resistance to the drug.

DETAILED DESCRIPTION:
ISIDE is a European, multicenter, open label, single-arm phase IIIB trial that aims to include 38 patients with pathologically documented locally advanced inoperable or metastatic triple negative breast cancer (mTNBC) whose disease has progressed on (neo)adjuvant chemotherapy with or without immunotherapy for early TNBC or within 6 months after the end of any systemic therapy, surgery or radiotherapy with curative intent, whatever comes last.

The primary objective is to to evaluate the efficacy of sacituzumab govitecan via investigator-assessed objective response rate (ORR) according to RECIST v1.1.

Patient will receive SG until disease progression, unacceptable toxicity, or decision to withdraw its participation.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have signed a written informed consent prior to any trial specific procedures;

   Note: When the patient is unable to write to give his written consent, a trusted person of their choice, independent from the investigator or the sponsor, can confirm in writing the patient's consent
2. Male or female ≥ 18 years of age;
3. Patients with pathologically documented locally advanced inoperable or metastatic triple negative breast cancer (mTNBC) whose disease has progressed on (neo)adjuvant chemotherapy+/-immunotherapy for early TNBC or within 6 months after the end of any systemic therapy, surgery or radiotherapy with curative intent, whatever comes last.

   Note: TNBC is defined as the absence of HER2 overexpression by immunohistochemistry (IHC) defined as IHC 0, 1+, or 2+ and fluorescence in situ hybridization [FISH] non-amplified and estrogen receptor (ER) expression <10% and progesterone receptor (PR) expression <10% by local pathological assessment on the most recent tissue sample collected
4. Prior exposure to a taxane

   Note: If indicated, prior therapy with ICI for patients with PD1 positive tumor and prior treatment with PARP inhibitor for patients with gBRCAm is required
5. Measurable disease, as defined by RECIST v1.1
6. Patient must have accepted to perform on-treatment biopsies. If the physician considers doing the biopsy on the primary tumor site because accessibility, it can be performed only if the primary tumor site has not been previously irradiated;
7. Have metastatic site easily accessible to biopsy (with exception of bone metastasis)

   Note 1: Patients with only bone metastasis will be eligible if the primary tumor is accessible for biopsy at inclusion

   Note 2: If the patient has a single measurable lesion and it is the only one that can be biopsied, the patient cannot be included because the disease is no longer measurable according to RECIST v1.1
8. Eastern Cooperative Oncology Group (ECOG) performance status ≤2;
9. Life expectancy ≥12 weeks;
10. Adequate haematologic and organ function
11. Negative hepatitis B surface antigen (HBsAg) test at screening (patients with a negative HBsAg test and a positive total hepatitis B core antibody (HBcAb) test at screening are eligible), negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening;
12. Evidence of post-menopausal status or negative pregnancy urinary test within 72 hours or serum pregnancy test within 14 days before study treatment and confirmed prior to treatment on Cycle 1 Day 1 for female pre-menopausal patients;
13. Woman of childbearing potential and male patient must agree to use adequate contraception for the duration of trial participation and up to 6 months after completing treatment for women and up to 3 months for men;
14. Patient affiliated to a social security system (or equivalent);
15. Patient is willing and able to comply with the protocol for the duration of the trial including undergoing treatment and scheduled visits, and examinations including follow-up;

Exclusion Criteria:

1. Participation in another therapeutic trial within the 30 days prior to C1D1;
2. Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases or evidence of leptomeningeal disease or clinically active spinal cord compression. Patients with stable and asymptomatic brain metastases will be eligible, yet the number will be capped to 15% of the overall population;
3. Previous history of cancer other than mTNBC within 5 years prior to C1D1, except of those with a negligible risk of metastasis or death (e.g., 5-year OS rate >90%) and treated with curative intent (e.g. carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or stage I uterine cancer);
4. Prior treatment with topoisomerase-1 inhibitor or with ADC containing topoisomerase-1 inhibitor
5. Met any of the following criteria for cardiac disease:

   1. Myocardial infarction or unstable angina pectoris within 6 months of enrolment.
   2. History of serious ventricular arrhythmia (ie, ventricular tachycardia or ventricular fibrillation), high-grade atrioventricular block, or other cardiac arrhythmias requiring antiarrhythmic medications (except for atrial fibrillation that is well controlled with antiarrhythmic medication); history of QT interval prolongation.
   3. New York Heart Association (NYHA) Class III or greater congestive heart failure or left ventricular ejection fraction of <40%.
6. Severe uncontrolled infection requiring oral or IV antibiotics within 4 weeks prior to C1D1;
7. Major surgical procedure within 4 weeks prior to C1D1;
8. History of severe allergic, anaphylactic, or other hypersensitivity reactions to humanized antibodies;
9. Known hypersensitivity to the study drug, its metabolites, or formulation excipient.
10. Patients receiving concomitant anti-cancer treatments such as chemotherapy, immunotherapy, endocrine therapy and radiotherapy;
11. Patients with unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved according to the common terminology criteria for adverse events of the National Cancer Institute (NCI-CTCAE) v5.0 grade >2
12. Treatment with systemic corticosteroids dosed at >20 mg prednisone or equivalent or other systemic immunosuppressive medications within 2 weeks prior to C1D1;
13. Known history of testing positive for HIV or known acquired immunodeficiency syndrome if not controlled;
14. Evidence of significant uncontrolled concomitant disease;
15. Requirement for ongoing therapy with medications that are prohibited or to be used with caution
16. Individuals with physical or psychological conditions considered not to be compatible with the trial;
17. Persons deprived of their liberty or under protective custody or guardianship;
18. Pregnant or breastfeeding women;
19. Patients unwilling or unable to comply with the medical follow-up required by the trial because of geographic, familial, social, or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2028-05-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | From inclusion to disease progression, up to 6 months
  ORR is defined as the number of patient with at least a confirmed complete response (CR) or partial response (PR), based on the best objective response values while on treatment

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From inclusion to disease progression or death, up to 2 years
  PFS iis the length of time during and after the treatment of a disease that a patient lives with the disease but it does not get worse.
Duration of response (DOR) | From inclusion to disease progression or death, up to 2 years
  DOR is defined as the time from the date of the first documentation of objective response (CR or PR) to the date of the first documentation of disease progression or death due to any cause
Clinical benefice risk (CBR) | From inclusion to disease progression or death, up to 2 years
  CBR is defined as the presence of at least a PR or CR, or a stable disease (SD) while on treatment
Overall Survival (OS) | From inclusion to disease progression or death, up to 2 years
  The overall survival is the length of time from randomization that patients enrolled in the study are still alive.
The incidence of adverse events (Safety) | Throughout study completion, up to 36 months
  Safety and tolerability of sacituzumab govitecan will be evaluated using the National Cancer Institute-Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5). NCI-CTCAE is widely accepted in the community of oncology research as the leading rating scale for adverse events. This scale, divided into 5 grades (1 = "mild", 2 = "moderate", 3 = "severe", 4 = "life-threatening", and 5 = "death") determined by the investigator, will make it possible to assess the severity of the disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Pistilli, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Gustave Roussy, Villejuif, France